CLINICAL TRIAL: NCT00000614
Title: Prevention of Recurrent Venous Thromboembolism (PREVENT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 117; R01HL057951 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Peripheral Vascular Diseases; Thromboembolism; Vascular Diseases; Venous Thromboembolism
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Peripheral Vascular Diseases; Thromboembolism; Vascular Diseases; Venous Thromboembolism | interventions — Warfarin

INTERVENTIONS:
Drug: warfarin

SUMMARY:
A multicenter randomized, double blind placebo controlled trial to determine the efficacy of long-term, low dose warfarin in the secondary prevention of venous thromboembolism.

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism is associated with more than 300,000 hospitalizations and results in thousands of deaths annually. Conventional therapy consists of intravenous heparin followed by oral anticoagulants usually given for three to six months. The recommended intensity of oral anticoagulants (warfarin) has been derived from clinical trials. Such therapy is usually quite effective. However, some patients develop recurrent disease after the oral anticoagulants are stopped. A recent randomized study evaluated the optimal duration of oral anticoagulant therapy. After acute treatment with heparin, subjects were treated with oral anticoagulants for either six weeks or six months with a target INR * of 2 to 2.85. There was no difference in mortality in the two groups. Recurrence was not seen while the patients were under treatment. When anticoagulants were stopped, recurrent thrombosis was documented in 18 percent of the patients treated for six weeks and in 9.5 percent of those treated for six months. The period of greatest risk of recurrence for the six weeks patients was immediately after therapy was stopped. There was a linear increase in cumulative risk of 5 to 6 percent per year for both treatment groups during the following 18 months.

For patients who have experienced idiopathic venous thrombosis, the risk of recurrence may continue even after several months of conventional therapy. Further prophylactic therapy might be beneficial for the patients who are at risk for late recurrence. But, because of the presumed risk of bleeding and inconvenience of monitoring standard warfarin therapy, most physicians usually limit treatment to three to six months.

In 1997, Simioni showed a cumulative recurrence rate of VTE of 39.7 percent among those with factor V Leiden mutation, with all recurrences occurring within three years, a rate 2.4 times higher than among individuals without the mutation. The factor V Leiden mutation is found in 4 to 6 percent of Caucasians and is the single most important cause of thromboembolism in a variety of conditions. Heterozygous carriers with the mutation have VTE at a younger age than do noncarriers. Among those with first VTE, the prevalence of the mutation is 15 to 40 percent and among those with a family history of VTE, as high as 50 percent. However, in a large study of men participating in the Physicians Health Study, those individuals with the mutation had an increased rate of VTE over time. These age-specific incidence rate differences ranged from 1.23 to 5.97 in those aged 70 or older. These data suggest that confounders other than genetic predisposition are important in the development of VTE.

* The INR or international normalized ratio is the ratio of patient prothrombin to control prothrombin multiplied by the international sensitivity index. The INR was introduced by the World Health Organization to standardize control of anticoagulant therapy internationally.

DESIGN NARRATIVE:

Multicenter, randomized, double-blind, placebo-controlled. A total of 253 patients were randomized to usual care plus placebo and a total of 255 patients to usual care plus a three-to-four year regimen of low-dose warfarin (target INR 1.5 to 2.0), which after initial titration required infrequent outpatient monitoring. Double-blind INR assessment and dose adjustment were performed every three months to ensure patient safety and to monitor compliance. Primary endpoints included recurrent venous thromboembolism, major bleeding episodes, and all-cause mortality. Separate analysis was performed of all-cause mortality in the total patient population and in those with factor V Leiden.

The study consisted of 52 clinical centers, a laboratory coordinating center, the clinical coordinating center, and the data coordinating center.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Patients with venous thromboembolism, including patients with factor V Leiden. Patients had completed prescribed anticoagulation therapy within the last two years before the trial and were not currently on anticoagulation therapy.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Glynn — Brigham and Women's Hospital

REFERENCES:
- [Background] Ridker PM. Long-term, low-dose warfarin among venous thrombosis patients with and without factor V Leiden mutation: rationale and design for the Prevention of Recurrent Venous Thromboembolism (PREVENT) trial. Vasc Med. 1998;3(1):67-73. doi: 10.1177/1358836X9800300114. PMID 9666536
- [Background] Ridker PM, Goldhaber SZ, Danielson E, Rosenberg Y, Eby CS, Deitcher SR, Cushman M, Moll S, Kessler CM, Elliott CG, Paulson R, Wong T, Bauer KA, Schwartz BA, Miletich JP, Bounameaux H, Glynn RJ; PREVENT Investigators. Long-term, low-intensity warfarin therapy for the prevention of recurrent venous thromboembolism. N Engl J Med. 2003 Apr 10;348(15):1425-34. doi: 10.1056/NEJMoa035029. Epub 2003 Feb 24. PMID 12601075
- [Background] Schafer AI. Warfarin for venous thromboembolism - walking the dosing tightrope. N Engl J Med. 2003 Apr 10;348(15):1478-80. doi: 10.1056/NEJMe030018. Epub 2003 Feb 24. No abstract available. PMID 12601074
- [Background] Miles JS, Miletich JP, Goldhaber SZ, Hennekens CH, Ridker PM. G20210A mutation in the prothrombin gene and the risk of recurrent venous thromboembolism. J Am Coll Cardiol. 2001 Jan;37(1):215-8. doi: 10.1016/s0735-1097(00)01080-9. PMID 11153741
- [Background] Sick PB, Brosteanu O, Ulrich M, Thiele H, Niebauer J, Busch I, Schuler G. Prospective randomized comparison of early and late results of a carbonized stent versus a high-grade stainless steel stent of identical design: the PREVENT Trial [corrected]. Am Heart J. 2005 Apr;149(4):681-8. doi: 10.1016/j.ahj.2004.07.011. PMID 15990753